CLINICAL TRIAL: NCT03590626
Title: Effect of Dulaglutide on Liver Fat in Patients With Type 2 Diabetes and Nonalcoholic Fatty Liver Disease: A Randomized Controlled Trial
Brief Title: Effect of Dulaglutide on Liver Fat in Patients With Type 2 Diabetes and Nonalcoholic Fatty Liver Disease
Acronym: D-LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medanta, The Medicity, India (Other)
Responsible Party: Principal Investigator, Dr Mohammad Shafi Kuchay, Consultant, Medanta, The Medicity, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMDLIFT01
Record Dates: First submitted 2018-06-11; First posted 2018-07-18 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Non Alcoholic Fatty Liver Disease; Type2 Diabetes Mellitus
Keywords: Non Alcoholic Fatty Liver Disease; Type 2 Diabetes Mellitus; GLP-1 receptor agonist; Dulaglutide; MRI-Proton density fat fraction; Fat Mapping; Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Intervention Model Description: will randomize the patients into either dulaglutide group or control group in a 1:1 ratio using computer-generated numbers
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dulaglutide group (Experimental): receive dulaglutide 0.75 mg weekly for 4 weeks followed by 1.5 mg weekly for 20 weeks plus standard treatment for type 2 diabetes
  Interventions: Drug: Dulaglutide
- Control group (No Intervention): receive standard treatment for type 2 diabetes and up titration of treatment will be done by anti-diabetic medicines other than the GLP-1 receptor agonist

INTERVENTIONS:
Drug: Dulaglutide — 0.75 mg weekly for 4 weeks followed by 1.5 mg weekly for 20 weeks
  Arms: Dulaglutide group

SUMMARY:
This D-LIFT (Effect of dulaglutide on Liver Fat) trial is an investigator initiated, prospective, open label, randomized clinical study to examine the effect of dulaglutide 0.75 mg subcutaneously weekly for 4 weeks, followed by 1.5 mg weekly for 20 weeks when included in the standard treatment for type 2 diabetes vs. standard treatment for type 2 diabetes (minus dulaglutide) in patients with type 2 diabetes and NAFLD. Hepatic steatosis (intracellular fat accumulation in hepatocytes) will be measured by MRI-PDFF, a validated quantitative biomarker for liver fat. The study will be conducted according to the CONSORT guidelines. The patient population for the trial will be derived from Medanta-The Medicity Hospital endocrine out-patient clinic, who would primarily visit for management of type 2 diabetes and other co-morbidities. The study will be conducted in Medanta-The Medicity Hospital, Gurugram, Haryana, which is a tertiary care center in North India. Patients deemed eligible will be screened for the trial. The clinical trial protocol will be presented for approval to the institutional ethics review board. Informed written consent will be obtained from all the participants before enrolment into the study.

DETAILED DESCRIPTION:
OBJECTIVE Nonalcoholic fatty liver disease (NAFLD) is a public health problem in patients with type 2 diabetes mellitus (T2DM). The presence of type 2 diabetes in patients with NAFLD is a risk factor for its progression to a more severe liver disease known as nonalcoholic steatohepatitis (NASH). NASH, in turn, can progress to liver fibrosis, cirrhosis and hepatocellular cancer in some patients. GLP-1 receptor agonists are a class of anti-diabetic agents that reduce hyperglycemia and body weight. Liraglutide is a daily injectable GLP-1 receptor agonist that has been shown to reduce liver fat in patients with type 2 diabetes and NAFLD. Dulaglutide is a weekly injectable GLP-1 receptor agonist that is approved for type 2 diabetes. Data regarding the effect of dulaglutide on liver fat are scarce. Therefore, the present study is planned to evaluate the effect of dulaglutide on liver fat in patients with type 2 diabetes and nonalcoholic fatty liver disease.

Materials and methods Study design This D-LIFT (Effect of dulaglutide on Liver Fat) trial is an investigator initiated, prospective, open label, randomized clinical study to examine the effect of dulaglutide 0.75 mg subcutaneously weekly for 4 weeks, followed by 1.5 mg weekly for 20 weeks when included in the standard treatment for type 2 diabetes vs. standard treatment for type 2 diabetes (minus dulaglutide) in patients with type 2 diabetes and NAFLD. Hepatic steatosis (intracellular fat accumulation in hepatocytes) will be measured by MRI-PDFF, a validated quantitative biomarker for liver fat. The study will be conducted according to the CONSORT guidelines. The patient population for the trial will be derived from Medanta-The Medicity Hospital endocrine out-patient clinic, who would primarily visit for management of type 2 diabetes and other co-morbidities. The study will be conducted in Medanta-The Medicity Hospital, Gurugram, Haryana, which is a tertiary care center in North India. Patients deemed eligible will be screened for the trial. The clinical trial protocol will be presented for approval to the institutional ethics review board. Informed written consent will be obtained from all the participants before enrolment into the study.

Inclusion and Exclusion Criteria

Patients will be enrolled in the study if they met all of the following criteria:

1. A man or woman, 20 years of age or above with the diagnosis of type 2 diabetes for at least 3 months who meets all of the following two criteria:

   1. On standard anti-diabetic agents (metformin, DPP-4 inhibitors, sulphonylureas or insulin, in any combination) with an HbA1c of ≤ 7.0% and ≥10.0% (≤53 and ≥86 mmol/mol) at screening
   2. Have documented hepatic steatosis (MRI-PDFF >6%) on screening MRI-PDFF
2. Subjects must be medically stable on the basis of medical history, physical examination and laboratory investigations.
3. Subjects must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
4. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of the study and are willing to participate in the study.

In addition, all the conditions described below will be considered exclusion criteria:

1. History of diabetic ketoacidosis, type 1 diabetes, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy.
2. History of brittle or labile glycemic control, with widely varying glucose measurements by FPG or SMBG such that stable glucose control over the treatment period would be unlikely.
3. History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 3 years before Screening, or an Alcohol Use Disorders Identification Test (AUDIT) with a score ≥8, or alcohol consumption of more than 20 g per day in the case of women and more than 30 g per day in the case of men for at least three consecutive months during the previous 5 years.
4. Thyroid stimulating hormone (TSH) value that is either < 0.45 mIU/L or >10 mIU/L at Screening.

   Note: Subjects on thyroid hormone replacement therapy must be on a stable dose and dosing regimen for at least 4 weeks prior to enrollment.
5. Use of a PPARγ agonist [e.g., a thiazolidinedione (pioglitazone], an SGLT2 inhibitor (e.g., canagliflozin, empagliflozin) or another GLP-1 receptor agonist (e.g., liraglutide) within 24 weeks before the enrollment.
6. BMI ≥23 kg/m2 or ≥40 kg/m2.
7. Ongoing eating disorder, or a significant weight loss or weight gain within 12 weeks before the Screening visit, defined as an increase or decrease of 5% in body weight based upon clinic-based measurement or, if not available, based on subject's report.
8. Use of weight loss medication (prescription and/or over-the-counter) within 3 months prior to Screening or have participated in a weight loss/diet program within 12 months prior to Screening.
9. Renal disease that required treatment with immunosuppressive therapy or a history of dialysis or renal transplant.
10. Myocardial infarction, unstable angina, pulmonary hypertension, revascularisation procedure (e.g., stent or bypass graft surgery), or cerebrovascular accident within 3 months before Screening, or revascularisation procedure is planned, or subject has a history of New York Heart Association (NYHA) Class III-IV cardiac disease.
11. History of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening.
12. Use of vitamin E within 3 months before screening.
13. History of prior bariatric (e.g., Roux-en-Y gastric bypass) or other major upper gastrointestinal surgical procedure (including gastric resection).
14. History of diabetic gastroparesis (or symptoms suggestive of this disorder, including postprandial bloating or vomiting), malabsorption, inflammatory bowel disease, or any other chronic, clinically important gastrointestinal disorder.
15. Estimated glomerular filtration rate (eGFR) <65 mL/min/1•73 m2 using the Modification of Diet in Renal Disease Study (MDRD) equation.
16. Subjects with a history of having or possibly having metallic material in the body or any contraindication for a MR examination.
17. Screening fasting serum triglycerides ≥600 mg/dL (6•74 mmol/L).
18. Claustrophobia, or anxiety related to previous negative experiences with magnetic resonance imaging procedures or if the subject is unwilling to participate in magnetic resonance imaging procedures.
19. Clinically important hematologic disorder (e.g., symptomatic anemia, proliferative bone marrow disorder, thrombocytopenia) at Screening.
20. History of human immunodeficiency virus (HIV) antibody positive at Screening.
21. Major surgery (e.g., requiring general anaesthesia) within 12 weeks before Screening, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study.
22. Contraindications to the use of dulaglutide (per DULAGLUTIDE US Prescribing Information).
23. Current use of a corticosteroid medication or immunosuppressive agent, or likely to require treatment with a corticosteroid medication or an immunosuppressive agent.

    Note: Subjects using inhaled, intranasal, intra-articular, or topical corticosteroids, or corticosteroids in therapeutic replacement doses may participate.
24. Pregnancy or women breastfeeding or planning to become pregnant while enroled in this study.
25. History of significant cardiac, vascular, pulmonary, renal, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances.
26. Use of drugs known to cause hepatic steatosis like methotrexate.

Baseline assessment at screening All patients will undergo a baseline assessment before randomization, including detailed medical history and physical examination.

Randomization A research assistant will randomize the patients into either dulaglutide group or control group in a 1:1 ratio using computer-generated numbers. SPSS software will be used to generate 60 random numbers between 000 to 999. The random numbers will be divided by 2 and the reminder noted. The reminders 0, & 1 will correspond to dulaglutide and control group respectively. It will be ensured that these are equal in number. Opaque envelopes will be prepared with serial number on the top and the assigned group inside the envelop. After recruiting the subjects, the envelop with corresponding serial number will be opened and the subjects assign to the relevant groups after opening the envelop. The patients will then be sent back to their respective consultants (MSK, SKM, KJF, AM) in the endocrine department for initiation and/or adjustment of treatment for type 2 diabetes (according to randomization into dulaglutide or control groups) and other co-morbidities. Treatment allocation will be open-label.

Study visits After careful assessment at the baseline visit, patients meeting all inclusion and exclusion criteria will be randomized to receive dulaglutide 0.75 mg weekly for 4 weeks followed by 1.5 mg weekly for 20 weeks plus standard treatment for type 2 diabetes. The control group will receive standard treatment for type 2 diabetes and up titration of treatment will be done by anti-diabetic medicines other than the GLP-1 receptor agonist. Patients will be advised to return to the out-patient endocrine clinic for follow-up visits at weeks 12 and 24.

Primary and secondary outcomes The primary outcome measure is change in liver fat quantified by MRI-PDFF in colocalized regions of interest (ROI) within each of the nine liver segments. The secondary outcome measures are change in serum AST, ALT and GGT values; Fibroscan, change in cardiometabolic markers namely IL-1, TNF-alpha, hs-CRP, leptin, adiponectin and homocysteine and fibrosis markers.

MRI-PDFF protocols MRI-PDFF for fat quantification MRI-PDFF is a non-invasive, objective, and quantitative MR imaging-based biomarker that can accurately estimate liver fat. MRI-PDFF has been demonstrated to be a robust technique for assessing treatment response in NASH clinical trials. In this study, the time interval from obtaining the baseline MRI-PDFF to initiating the study drug will be less than one week.

MRI-PDFF for detailed fat mapping of the entire liver All MR examinations will be done by an experienced MR technologist in the Medanta Radiology department under the direction of the radiologist investigator (SK). The radiologist investigator, blinded to the patients' treatment group allocation, clinical and biochemical data, and order of scans (baseline and follow-up), will perform the image analyses.

ROI colocalization before and after treatment To assess longitudinal changes in liver fat content, one colocalized ROI will be placed in each of the nine liver segments (nine separate ROIs) on the baseline and follow-up MRI examinations.

Statistical analysis Plan The analysis will include profiling of patients on different demographic, clinical and laboratory parameters etc. Quantitative data will be presented in terms of means and standard deviation and qualitative/categorical data will be presented as absolute numbers and proportions. To compare between the two groups, the Chi-squared test or Fisher's exact test will be used for categorical variables, and the independent samples t test or Wilcoxon-Mann-Whitney U test will be used for the differences between continuous variables. Pearson correlation coefficient will be used to evaluate correlations between variables. Additional analyses of primary and secondary outcomes within treatment groups will be performed by using two-tailed independent sample t tests, paired t tests, or non-parametric tests, when indicated. P-value < 0.05 is considered statistically significant. SPSS software will be used for analysis.

Sample size calculation Investigator assumed that a 5% difference between dulaglutide and control groups would be the minimally appreciable and clinically relevant difference. Based on the results of previous similar clinical studies involving colesevelam and ezetimibe, Investigatorexpected the empagliflozin group to have a liver fat reduction of >5% compared to baseline, the control group to have <1% reduction in liver fat compared to baseline, and a dropout rate of <10%. With these assumptions the sample size per group works out as ≥20 to achieve a power of at least 90% with a β of 0.05. Therefore, Investigator plan to randomize 60 patents, 30 in each group to ensure adequate study power even with dropouts.

Method of sample size calculation

Assumptions:

Change in liver fat from baseline to week 20 in dulaglutide group (m1) = 5.0 unit Change in liver fat from baseline to week 20 in control group (m2) = 1.0 unit Confidence level -95% Power - 90% Coefficient of variation = 80%

Formula for sample size calculation:

n = (Zα+Zβ)2 * (σ12 + σ22)) / (m1-m2)2, where Zα is the value of normal distribution corresponding to desired confidence level Zβ is the value of the Normal distribution corresponding to desired power σ1 and σ2 are the standard deviation of the two groups With these assumptions the sample size per group works out as 20. Investigator will randomize 30 in each group to ensure adequate power even after dropouts.

Patient confidentiality Precautions will be taken to ensure confidentiality. Data collection forms will not reveal the name of patients included in study. All the participants will be covered by insurance to cover the cost of any untoward effect directly resulting from enrolment in the study.

ELIGIBILITY:
Inclusion Criteria:

1. A man or woman, 20 years of age or above with the diagnosis of type 2 diabetes for at least 3 months who meets all of the following two criteria:

   1. On standard anti-diabetic agents (metformin, DPP-4 inhibitors, sulphonylureas or insulin, in any combination) with an HbA1c of ≤ 7.0% and ≥10.0% (≤53 and ≥86 mmol/mol) at screening
   2. Have documented hepatic steatosis (MRI-PDFF >6%) on screening MRI-PDFF
2. Subjects must be medically stable on the basis of medical history, physical examination and laboratory investigations.
3. Subjects must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
4. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of the study and are willing to participate in the study

Exclusion Criteria:

1. History of diabetic ketoacidosis, type 1 diabetes, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy.
2. History of brittle or labile glycemic control, with widely varying glucose measurements by FPG or SMBG such that stable glucose control over the treatment period would be unlikely.
3. History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 3 years before Screening, or an Alcohol Use Disorders Identification Test (AUDIT) with a score ≥8, or alcohol consumption of more than 20 g per day in the case of women and more than 30 g per day in the case of men for at least three consecutive months during the previous 5 years.
4. Thyroid stimulating hormone (TSH) value that is either < 0.45 mIU/L or >10 mIU/L at Screening.

   Note: Subjects on thyroid hormone replacement therapy must be on a stable dose and dosing regimen for at least 4 weeks prior to enrollment.
5. Use of a PPARγ agonist [e.g., a thiazolidinedione (pioglitazone], an SGLT2 inhibitor (e.g., canagliflozin, empagliflozin) or another GLP-1 receptor agonist (e.g., liraglutide) within 24 weeks before the enrollment.
6. BMI ≥23 kg/m2 or ≤40 kg/m2.
7. Ongoing eating disorder, or a significant weight loss or weight gain within 12 weeks before the Screening visit, defined as an increase or decrease of 5% in body weight based upon clinic-based measurement or, if not available, based on subject's report.
8. Use of weight loss medication (prescription and/or over-the-counter) within 3 months prior to Screening or have participated in a weight loss/diet program within 12 months prior to Screening.
9. Renal disease that required treatment with immunosuppressive therapy or a history of dialysis or renal transplant.
10. Myocardial infarction, unstable angina, pulmonary hypertension, revascularisation procedure (e.g., stent or bypass graft surgery), or cerebrovascular accident within 3 months before Screening, or revascularisation procedure is planned, or subject has a history of New York Heart Association (NYHA) Class III-IV cardiac disease.
11. History of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening.
12. Use of vitamin E within 3 months before screening.
13. History of prior bariatric (e.g., Roux-en-Y gastric bypass) or other major upper gastrointestinal surgical procedure (including gastric resection).
14. History of diabetic gastroparesis (or symptoms suggestive of this disorder, including postprandial bloating or vomiting), malabsorption, inflammatory bowel disease, or any other chronic, clinically important gastrointestinal disorder.
15. Estimated glomerular filtration rate (eGFR) <65 mL/min/1•73 m2 using the Modification of Diet in Renal Disease Study (MDRD) equation.
16. Subjects with a history of having or possibly having metallic material in the body or any contraindication for a MR examination.
17. Screening fasting serum triglycerides ≥600 mg/dL (6•74 mmol/L).
18. Claustrophobia, or anxiety related to previous negative experiences with magnetic resonance imaging procedures or if the subject is unwilling to participate in magnetic resonance imaging procedures.
19. Clinically important hematologic disorder (e.g., symptomatic anemia, proliferative bone marrow disorder, thrombocytopenia) at Screening.
20. History of human immunodeficiency virus (HIV) antibody positive at Screening.
21. Major surgery (e.g., requiring general anaesthesia) within 12 weeks before Screening, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study.
22. Contraindications to the use of dulaglutide (per DULAGLUTIDE US Prescribing Information).
23. Current use of a corticosteroid medication or immunosuppressive agent, or likely to require treatment with a corticosteroid medication or an immunosuppressive agent.

    Note: Subjects using inhaled, intranasal, intra-articular, or topical corticosteroids, or corticosteroids in therapeutic replacement doses may participate.
24. Pregnancy or women breastfeeding or planning to become pregnant while enroled in this study.
25. History of significant cardiac, vascular, pulmonary, renal, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances.
26. Use of drugs known to cause hepatic steatosis like methotrexate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Change in liver fat | Baseline to 24 weeks
  change in liver fat quantified by MRI-PDFF in colocalized regions of interest (ROI) within each of the nine liver segments

SECONDARY OUTCOMES:
Change in Biochemical Markers | Basline to 24 weeks
  change in serum AST levels
Change in Fibroscan Parameters | Basline to 24 weeks
  Change in liver stiffness measurement (LSM) in kPa
Change in Fibroscan Parameters | Basline to 24 weeks
  Change in Controlled Attenuation Parameter (CAP) in dB/m
change in cardiometabolic markers | Basline to 24 weeks
  change in cardiometabolic markers namely IL-1, TNF-alpha, hs-CRP, leptin, adiponectin and homocysteine and fibrosis markers
Change in Biochemical Markers | Baseline to 24 weeks
  Change in serum ALT levels
Change in Biochemical Markers | Baseline to 24 weeks
  change in serum GGT levels

CONTACTS AND LOCATIONS:
Locations (1):
- Division Of Endocrinology & Diabetes, Medanta The Medicity, Gurgaon, Haryana, India

REFERENCES:
- [Background] Umpierrez G, Tofe Povedano S, Perez Manghi F, Shurzinske L, Pechtner V. Efficacy and safety of dulaglutide monotherapy versus metformin in type 2 diabetes in a randomized controlled trial (AWARD-3). Diabetes Care. 2014 Aug;37(8):2168-76. doi: 10.2337/dc13-2759. Epub 2014 May 19. PMID 24842985
- [Result] Bouchi R, Nakano Y, Fukuda T, Takeuchi T, Murakami M, Minami I, Izumiyama H, Hashimoto K, Yoshimoto T, Ogawa Y. Reduction of visceral fat by liraglutide is associated with ameliorations of hepatic steatosis, albuminuria, and micro-inflammation in type 2 diabetic patients with insulin treatment: a randomized control trial. Endocr J. 2017 Mar 31;64(3):269-281. doi: 10.1507/endocrj.EJ16-0449. Epub 2016 Dec 3. PMID 27916783
- [Result] Petit JM, Cercueil JP, Loffroy R, Denimal D, Bouillet B, Fourmont C, Chevallier O, Duvillard L, Verges B. Effect of Liraglutide Therapy on Liver Fat Content in Patients With Inadequately Controlled Type 2 Diabetes: The Lira-NAFLD Study. J Clin Endocrinol Metab. 2017 Feb 1;102(2):407-415. doi: 10.1210/jc.2016-2775. PMID 27732328
- [Result] Dungan KM, Povedano ST, Forst T, Gonzalez JG, Atisso C, Sealls W, Fahrbach JL. Once-weekly dulaglutide versus once-daily liraglutide in metformin-treated patients with type 2 diabetes (AWARD-6): a randomised, open-label, phase 3, non-inferiority trial. Lancet. 2014 Oct 11;384(9951):1349-57. doi: 10.1016/S0140-6736(14)60976-4. Epub 2014 Jul 10. PMID 25018121
- [Result] Nauck M, Weinstock RS, Umpierrez GE, Guerci B, Skrivanek Z, Milicevic Z. Efficacy and safety of dulaglutide versus sitagliptin after 52 weeks in type 2 diabetes in a randomized controlled trial (AWARD-5). Diabetes Care. 2014 Aug;37(8):2149-58. doi: 10.2337/dc13-2761. Epub 2014 Apr 17. PMID 24742660
- [Result] Giorgino F, Benroubi M, Sun JH, Zimmermann AG, Pechtner V. Efficacy and Safety of Once-Weekly Dulaglutide Versus Insulin Glargine in Patients With Type 2 Diabetes on Metformin and Glimepiride (AWARD-2). Diabetes Care. 2015 Dec;38(12):2241-9. doi: 10.2337/dc14-1625. Epub 2015 Jun 18. PMID 26089386
- [Result] Patel NS, Peterson MR, Brenner DA, Heba E, Sirlin C, Loomba R. Association between novel MRI-estimated pancreatic fat and liver histology-determined steatosis and fibrosis in non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2013 Mar;37(6):630-9. doi: 10.1111/apt.12237. Epub 2013 Feb 5. PMID 23383649
- [Result] Reeder SB, Cruite I, Hamilton G, Sirlin CB. Quantitative Assessment of Liver Fat with Magnetic Resonance Imaging and Spectroscopy. J Magn Reson Imaging. 2011 Oct;34(4):729-749. doi: 10.1002/jmri.22775. Epub 2011 Sep 16. PMID 22025886
- [Result] Permutt Z, Le TA, Peterson MR, Seki E, Brenner DA, Sirlin C, Loomba R. Correlation between liver histology and novel magnetic resonance imaging in adult patients with non-alcoholic fatty liver disease - MRI accurately quantifies hepatic steatosis in NAFLD. Aliment Pharmacol Ther. 2012 Jul;36(1):22-9. doi: 10.1111/j.1365-2036.2012.05121.x. Epub 2012 May 3. PMID 22554256
- [Result] Le TA, Chen J, Changchien C, Peterson MR, Kono Y, Patton H, Cohen BL, Brenner D, Sirlin C, Loomba R; San Diego Integrated NAFLD Research Consortium (SINC). Effect of colesevelam on liver fat quantified by magnetic resonance in nonalcoholic steatohepatitis: a randomized controlled trial. Hepatology. 2012 Sep;56(3):922-32. doi: 10.1002/hep.25731. Epub 2012 Jul 2. PMID 22431131
- [Result] Loomba R, Sirlin CB, Ang B, Bettencourt R, Jain R, Salotti J, Soaft L, Hooker J, Kono Y, Bhatt A, Hernandez L, Nguyen P, Noureddin M, Haufe W, Hooker C, Yin M, Ehman R, Lin GY, Valasek MA, Brenner DA, Richards L; San Diego Integrated NAFLD Research Consortium (SINC). Ezetimibe for the treatment of nonalcoholic steatohepatitis: assessment by novel magnetic resonance imaging and magnetic resonance elastography in a randomized trial (MOZART trial). Hepatology. 2015 Apr;61(4):1239-50. doi: 10.1002/hep.27647. Epub 2015 Feb 27. PMID 25482832
- [Derived] Kuchay MS, Krishan S, Mishra SK, Choudhary NS, Singh MK, Wasir JS, Kaur P, Gill HK, Bano T, Farooqui KJ, Mithal A. Effect of dulaglutide on liver fat in patients with type 2 diabetes and NAFLD: randomised controlled trial (D-LIFT trial). Diabetologia. 2020 Nov;63(11):2434-2445. doi: 10.1007/s00125-020-05265-7. Epub 2020 Aug 31. PMID 32865597